CLINICAL TRIAL: NCT06985719
Title: Effectiveness of Adapted Physical Activity Programs in Preventing Falls in People Aged Over 65: a Prospective Multicenter Study Carried Out Within the Maisons Sport Santé of Ile de France Departement
Brief Title: Effectiveness of Adapted Physical Activity Programs in Preventing Falls in People Aged Over 65
Acronym: APA-SAFE
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Médical Porte Verte (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-A00460-49
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-02

CONDITIONS: Adapted Physical Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to evaluate the effectiveness of Adapted Physical Activity (APA) programs offered by Sport-Health Centers (MSS) in reducing the risk of falls in the elderly.

DETAILED DESCRIPTION:
The effectiveness of adapted physical activity in preventing falls will be assessed by the evolution of SPPB before and after APA.

Evaluate the impact of APA on physical tests such as the UGT, the single-legged support test, to predict the risk of falling.

- Evaluate the impact of APA on risk factors associated with the risk of falling, such as fear of falling, overall perception of one's health, and depression.

All tests will be assessed at baseline and at the final visit 3 months after APA

ELIGIBILITY:
Inclusion Criteria:

* People at risk of falling People practicing an APA program for 3 months Persons who have given their consent to participate in the study

Exclusion Criteria:

* Patient refusal to participate in the study Absolute or relative contraindication to APA Persons under guardianship Non-affiliation to a social security scheme

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: This study aims to target people aged over 65, considered to be at risk of falling.
  Several methods have been validated in the existing literature to screen these patients. The chosen method is the Global Guide for Falls Prevention
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
SPPB Short Physical Performance Battery | Twice throughout study at baseline and 3 months after intervention
  This composite score is based on three tests: a balance test, a walking speed test, and the chair rise test